CLINICAL TRIAL: NCT03949582
Title: A Double-Blind Randomised Controlled Trial Investigating the Acute Effects of Mycoprotein on Glycaemic Control and Appetite in South Asian and Caucasian Adults With Type 2 Diabetes Mellitus
Brief Title: Acute Mycoprotein Effect on Glycaemic Control in South Asians
Acronym: ACMYCO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 18HH4870
Record Dates: First submitted 2019-05-08; First posted 2019-05-14 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes; South Asian; Guar gum; Mycoprotein; Caucasian; Glycaemic control; Appetite
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Double-Blind Crossover Randomised Controlled Trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mycoprotein as in Soup (Experimental): 24 will be randomised to soup (12 caucasian and 12 south asian) in order to test raw mycoprotein. Test food will be administrated orally and allowed 15 minutes for consumption at an even pace.
  Interventions: Other: Test food containing different types of dietary protein
- Mycoprotein as in Mince (Experimental): 24 will be randomised to mince (12 caucasian and 12 south asian) in order to test processed mycoprotein (Quorn). Test food will be administrated orally and allowed 15 minutes for consumption at an even pace.
  Interventions: Other: Test food containing different types of dietary protein

INTERVENTIONS:
Other: Test food containing different types of dietary protein — The test foods will be (in six study visits):
  Soy mince/soup Chicken mince/soup Quorn mince/soup Soy mince/soup with guar gum Chicken mince/soup with guar gum Quorn mince/soup with guar gum

SUMMARY:
Diet is the cornerstone treatment to manage blood sugar in people with Type 2 Diabetes (T2D). Fibres like guar gum and protein are macronutrients that have an effect in blood sugar levels. Mycoprotein is a fungi-based food high in both dietary fibre and protein shown to have a role in regulating blood sugar levels in healthy. However, little is known about the effects of mycoprotein on blood sugar levels in people with T2D. We are interested in South Asian because they have a different blood sugar response to the same food than a Caucasian.

The main aims of the study is to assess:

* The effect of mycoprotein in different formats (soup or mince) in blood sugar levels and appetite in South Asian and Caucasian with Type 2 Diabetes.
* The effect of the combination of mycoprotein with guar gum in different formats (soup or mince) in blood sugar levels and appetite in South Asian and Caucasian with T2D.

DETAILED DESCRIPTION:
This is a double-blind crossover RCT. A total of 48 participants (24 Caucasian and 24 South Asian) with T2D and non insulin treated will be recruited. Participant will be randomly allocated to one of these two groups:

Group 1: Test food in form of soup and Group 2: Test food in form of mince. Once allocated in one of the groups, participant will consume in a random order 6 different test foods (soy, chicken, mycoprotein with and without guar gum) in a determined format (either as in soup or mince).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Type 2 Diabetes Mellitus without insulin treatment.
* South Asian (Afghanistan, Bangladesh, Bhutan, Maldives, Nepal, India, Pakistan and Sri Lanka) or Caucasian Ancestry.
* Age 18-70
* 5.5% ≤ HbA1c ≤ 9.0%
* BMI ≤ 35.0
* If anti-diabetic regime or lipid lowering drugs are used, they have to be stable and controlled for at least 2 months; regimes are expected to remain stable throughout the duration of the study or not being on anti-diabetic medication.
* If on oral hypoglycaemic agent, participant should have the last dose at 8pm of the day before each study visit.
* Willingness to comply with the study protocol, including:
* Use of standard evening meal the day prior to the assessments
* Refrain from alcohol consumption (24 h prior the visit) and extraneous physical exercise (72 h prior to and during the assessments).
* Not changing physical activity routine or dietary habits for the duration of the study (except from the standard evening meal).

Exclusion Criteria:

* Not diagnosed with Type 2 Diabetes Mellitus
* Mixed ancestors
* Taking any of the following medications:
* Insulin
* Diabetic medication (except from Metformin or oral hypoglycaemic which are allowed).
* Orlistat
* Any gastrointestinal disease that interferes with bowel function and nutritional intake (i.e. Diabetes related constipation or diarrhoea secondary to neuropathy or chronic inflammatory bowel disease, gastrectomy, etc.)
* Significant heart (New York Heart Association class IV), hepatic (transaminase levels greater than 3 times normal) or renal disease (requiring dialysis)
* Cancer
* Pancreatitis
* Major infections (requiring antibiotics) within 3 weeks before study entry
* Concomitant therapy with acarbose, meglitinides, insulin, systemic glucocorticoids or within 2 weeks prior to study entry
* History of alcohol and/or drug abuse
* Investigator's uncertainty about the willingness or ability of patient to comply with the protocol requirements
* Participation in other nutrition trials within 3 months of study entry or drug trials within 5 months of study end
* Current smokers
* Allergic to test food or traces contained in the test food, breathing mould, penicillin, egg, soy
* Asthmatics.
* Any condition involving the imbalance of hormones
* Hypothyroidism.
* Weight change of ≥ 5% in the preceding 3 months
* Shift workers
* Vegetarian
* Medical implants that require batteries such as heart pace makers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Blood glucose | 180 minutes
  Fasting and Postprandial blood glucose
Blood insulin | 180 minutes
  Fasting and Postprandial blood insulin

SECONDARY OUTCOMES:
Subjective appetite feelings | 180 minutes
  Measured using Visual Analogue Scale from 0 to 100 milimetres, being 100 milimetres the higher score.
  Questions assessed are:
  1. "how hungry do you feel?"
  2. "how sick do you feel?"
  3. "how strong is your desire to eat?"
  4. "how much food do you think you could eat?"
  5. "how full do you feel?"
  6. "what is your level of satiety?"
  For questions 1 to 4 the desirable outcome considered as "good result" for the test food mycoprotein are values less than 30 milimetres, and for questions 5 and 6, values above 60 milimetres.
Ad libitum energy intake | At timepoint 180 minutes
  Measured using a buffet meal composed of wihte pasta with tomato sauce and weighting the serving bowl before and after to measure consumed grams of food.
Energy intake 72 hours post study visit | For 3 days after study visit
  Energy intake of free-living subjects will be measured using self reported food diaries

CONTACTS AND LOCATIONS:
Overall Officials: Gary Frost, Principal Investigator — Imperial College London
Locations (1):
- NIHR Imperial Clinical Research Facility, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No